CLINICAL TRIAL: NCT04236739
Title: Randomized Controlled Trial Comparing Clinical Outcomes of Instant MSC Product Accompanying Autologous Chondron Transplantation (IMPACT) for Focal Articular Cartilage Lesions of the Knee to Conservative Treatment
Brief Title: Comparing Clinical Outcomes of the One-step Cartilage Transplantation in Cartilage Defects of the Knee With Conservative Treatment
Acronym: IMPACT2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: R.J.H. Custers (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, R.J.H. Custers, Principal Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-455; NL67161.000.18 (Registry Identifier: CCMO); 2018-003470-27 (EudraCT Number)
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Cartilage Damage
Keywords: Cartilage; Cartilage damage; Cell therapy; MSC; ATMP; Knee; IMPACT; ACI; Chondrons
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. At baseline, participants will be randomized with variable block randomisation method to either group A in which case they receive IMPACT-treatment, or group B that will receive standard care. Standard care consists of optional physical therapy and pain medication. After 9 months, participants in group B can receive the intervention as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMPACT (Experimental): Application of a mixture of allogenic MSC's and autologous chondrons with a fibrin cell carrier (Tisseel®) during one surgical procedure.
  Interventions: Drug: Instant MSC Product accompanying Autologous Chondron Transplantation
- Control (No Intervention): Optional physical therapy or pain medication, according to participants' desire for 9 months.

INTERVENTIONS:
Drug: Instant MSC Product accompanying Autologous Chondron Transplantation — Application of a mixture of allogenic MSC's and autologous chondrons with a fibrin cell carrier (Tisseel®) in the cartilage defect of the knee during one surgical procedure.
  Arms: IMPACT

SUMMARY:
Articular cartilage defects in the knee have poor intrinsic healing capacity and may lead to functional disability and osteoarthritis. Cartilage cell therapy using autologous chondrocyte implantation has been established as the first advanced treatment therapy medicinal product. Although this technique has achieved good mid-term results, it is a costly and extensive two-stage procedure. 'Instant MSC Product accompanying Autologous Chondron Transplantation' (IMPACT) combines autologous recycled chondrons (chondrocytes surrounded by pericellular matrix) with MSCs for one-stage treatment of cartilage defects. IMPACT was successfully executed in a first-in-man phase I/II clinical trial in which 35 participants with cartilage defects were treated. The results showed a good safety profile, proper feasibility and good initial clinical efficacy at 18 months follow-up. Also good outcome at 24 and 36 months was shown in ongoing post study surveying of the participants. Consequently a new study with IMPACT was designed; IMPACT2. The objective of IMPACT2 is to compare clinical outcomes of 30 individual participants with cartilage defects treated with IMPACT to 30 participants treated with standard care for 9 months (consisting of optional physical therapy and pain medication). Participants should be aged 18-45 years with a symptomatic Modified Outerbridge Grade III or IV cartilage lesion of the knee ranging in size 2-8 cm^2.

After enrolment, participants will be allocated (randomized) to either group A in which case they receive IMPACT-treatment, or group B that will receive standard care. Standard care consists of optional physical therapy and pain medication. After 9 months, participants in group B can receive the IMPACT-procedure as well.

DETAILED DESCRIPTION:
IMPACT is designed as a one-stage cell-based regenerative therapy for isolated articular cartilage lesions. The investigational product consists of two cell types. Firstly, allogeneic MSCs, which are an "off-the-shelf" ATMP and also being used in a clinical trial for the treatment of steroid-resistant Graft versus Host Disease. Secondly, defect derived autologous chondrons that are reinserted into the defect in combination with MSCs within one procedure. During surgery, the autologous defect derived chondrons will be combined with allogeneic cryopreserved and thawed MSCs to enhance cartilage formation. Cells will be combined at a ratio of 10% chondrons and 90% MSCs and mixed in Tisseel® which will act as a cell carrier scaffold. In the phase I-II trial we showed no significant differences in clinical outcome between these dosages. Tisseel® is a registered widely used two-component adhesive containing fibrinogen and thrombin concentrate. When mixed, these components mimic the final steps of blood coagulation and form a stable physiological fibrin clot. The ATMP will be applied to the cartilage defect in a concentration of approximately 2 million cells per ml of fibrin glue, 0,5 to 0,7 ml per cm^2 will be administered. The amount of MSCs and chondrons is thus dependant of the size of the lesion. The cells will be applied in a ratio of 10:90 autologous chondrons: allogeneic MSCs.

To evaluate the clinical status/ improvement of the participants treated with the IMPACT therapy, the included participants will be asked to complete the Knee injury and Osteoarthritis Outcome Scoring (KOOS) and the EuroQoL 5-Dimension Health Questionnaire (EQ5D) at baseline (before IMPACT therapy) and at 3, 6, 9, 12 and 18 months follow-up.

To evaluate work leave and medical consumption a modified version iMTA Productivity cost questionnaire and iMTA Medical Consumption Questionnaire will be used.

A cost-effectiveness analysis will be performed to evaluate the extent to which IMPACT therapy affects costs compared to current treatment techniques. The costs of the procedures that are performed (i.e. IMPACT or current practice), as well as the costs of the product that is used (materials, operation theatre etc.), and the duration of the accompanying hospitalization episode, will be determined using the UMC Utrecht administrative data and study budget. In addition, the results of the iMTA Medical Consumption Questionnaire and the iMTA Productivity cost questionnaire will be used to collect data on respectively resource use and productivity loss during the rehabilitation period. All resource use will be multiplied with cost prizes, which will be obtained from the Dutch Healthcare Authority or from the Dutch manual for performing health economic evaluations, to calculate total societal costs. These costs will be combined with the QoL outcome measures (as described previously), to obtain an estimate of the cost-effectiveness of IMPACT as compared to current practice.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be eligible for the study:

* Provides written informed consent, is able to understand the content of the study, understands the requirements for follow-up visits and is willing to provide the required information at follow-up visits and in the questionnaires.
* Symptomatic articular cartilage lesion of the knee (femoral condyles or trochlea).
* Age >18 and <45 years old

Inclusion criteria during surgery

* Participants must meet the following secondary criteria to be eligible for the study:
* Modified Outerbridge Grade III or IV isolated cartilage lesion of the knee.
* A post-debridement size of the cartilage lesion > 2cm2 and ≤ 8 cm2
* At least 50% of functional meniscus remaining. Meniscal repair or resection is allowed during the IMPACT surgery provided that the surgeon is able to confirm that at least 50% of functional meniscus remains.
* Stable knee ligaments (i.e. anterior and posterior cruciate ligaments).

Exclusion Criteria:

* Malalignment of >5 degrees
* (History of) osteoarthritis, defined as Kellgren-Lawrence grade >3 as determined from appropriate X-ray.
* Concomitant inflammatory disease that affects the joint (rheumatoid arthritis, metabolic bone disease, psoriasis, gout, symptomatic chondrocalcinosis)
* (History of) Septic arthritis.
* (History of) Total meniscectomy in the target knee joint.
* Any surgery in the knee joint 6 months prior to study inclusion.
* Risk groups for MRI scanning due to the magnetic field like participants with pacemakers, nerve stimulators, metal particles, stents, clips or implants, (possible) pregnancy or breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical change on scale of 0-100 | At baseline, 3, 6 and 9 months
  KOOS-questionnaire (Knee injury and Osteoarthritis Outcome Score, 100 indicating no symptoms and 0 indicating extreme symptoms)
Quality of life change on scale of 0-100 | At baseline, 3, 6 and 9 months
  EQ-5d-questionnaire (The EQ-5D-5L has 5 dimensions, each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.)

SECONDARY OUTCOMES:
Structural change of the cartilage tissue | At baseline, 6 and 18 months
  MRI-scan

OTHER OUTCOMES:
Change in healtcare use and costs | At baseline, 3, 6, 9, 12 and 18 months
  iMTA-questionnaire (Medical Consumption and Productivity Cost Questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] de Windt TS, Vonk LA, Slaper-Cortenbach IC, van den Broek MP, Nizak R, van Rijen MH, de Weger RA, Dhert WJ, Saris DB. Allogeneic Mesenchymal Stem Cells Stimulate Cartilage Regeneration and Are Safe for Single-Stage Cartilage Repair in Humans upon Mixture with Recycled Autologous Chondrons. Stem Cells. 2017 Jan;35(1):256-264. doi: 10.1002/stem.2475. Epub 2016 Aug 29. PMID 27507787
- [Background] de Windt TS, Vonk LA, Slaper-Cortenbach ICM, Nizak R, van Rijen MHP, Saris DBF. Allogeneic MSCs and Recycled Autologous Chondrons Mixed in a One-Stage Cartilage Cell Transplantion: A First-in-Man Trial in 35 Patients. Stem Cells. 2017 Aug;35(8):1984-1993. doi: 10.1002/stem.2657. Epub 2017 Jun 23. PMID 28600828
- [Background] Korpershoek JV, Vonk LA, Kester EC, Creemers LB, de Windt TS, Kip MMA, Saris DBF, Custers RJH. Efficacy of one-stage cartilage repair using allogeneic mesenchymal stromal cells and autologous chondron transplantation (IMPACT) compared to nonsurgical treatment for focal articular cartilage lesions of the knee: study protocol for a crossover randomized controlled trial. Trials. 2020 Oct 9;21(1):842. doi: 10.1186/s13063-020-04771-8. PMID 33036661
- [Background] Saris TFF, de Windt TS, Kester EC, Vonk LA, Custers RJH, Saris DBF. Five-Year Outcome of 1-Stage Cell-Based Cartilage Repair Using Recycled Autologous Chondrons and Allogenic Mesenchymal Stromal Cells: A First-in-Human Clinical Trial. Am J Sports Med. 2021 Mar;49(4):941-947. doi: 10.1177/0363546520988069. Epub 2021 Feb 16. PMID 33591794